CLINICAL TRIAL: NCT07125937
Title: ROLE OF SILVER DIAMINE FLUORIDE (SDF) IN ARRESTING ENAMEL CARIES IN ADULTS REPORTING TO DENTAL COLLEGE HITEC-IMS TAXILA
Brief Title: Silver Diamine Flouride in Arresting Enamel Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Kinza Iftikhar, Kinza Iftikhar, HITEC-Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dr Kinza
Record Dates: First submitted 2025-08-11; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Carious Lesion
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 38% Silver Diamine Fluoride Application (Experimental): Participants will receive a single application of 38% Silver Diamine Fluoride (Advantage Arrest™, Elevate Oral Care LLC) on enamel caries lesions (ICDAS scores 1-3) in molars and premolars, following the UCSF protocol. Lesions will be evaluated clinically (ICDAS) and radiographically (ICCMS) at 3 weeks and 3 months post-treatment to assess caries arrest.
  Interventions: Drug: 38% Silver Diamine Fluoride

INTERVENTIONS:
Drug: 38% Silver Diamine Fluoride — A topical ammonia solution containing silver and fluoride ions applied directly to enamel caries lesions. Application will follow the UCSF protocol: lesions will be cleaned, isolated, and treated with SDF for 2 minutes using a microbrush applicator.

SUMMARY:
This interventional study aims to evaluate the effectiveness of 38% Silver Diamine Fluoride (SDF) in arresting enamel caries in adults aged 18-50 years. Dental caries is a biofilm-mediated, multifactorial disease that can cause progressive tooth damage. Conventional treatments are invasive and costly, whereas SDF offers a non-invasive, low-cost alternative. A total of 250 patients meeting the inclusion criteria will be treated with SDF following the UCSF protocol. Lesions will be evaluated clinically using ICDAS and radiographically using ICCMS at 3 weeks and 3 months post-intervention. The primary outcome is the proportion of enamel caries lesions arrested after treatment. Data will be analyzed using the chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Age group of subjects between 18 - 50 years

Carious lesions with ICDAS score 1, 2 and 3 in molars and premolars

Exclusion Criteria:

* PDL widening with periapical radiolucency around molars and premolars

Premolars and Molars with any white lesions other than caries

Third molars

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Proportion of enamel caries lesions arrested after SDF application | 3 months post-intervention
  Lesions will be clinically evaluated using the International Caries Detection and Assessment System (ICDAS) and radiographically using the International Caries Classification and Management System (ICCMS). Arrest is defined as no progression in ICDAS score and no radiographic progression

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kinza Iftikhar, BDS, Principal Investigator — HITEC-Institute of Medical Sciences
Locations (1):
- Hitec Ims, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33347946/